CLINICAL TRIAL: NCT00017680
Title: Study of High-Dose Melphalan and Autologous Stem Cell Transplantation in
Brief Title: Study of High-Dose Melphalan and Autologous Stem Cell Transplantation in Patients With Primary Light Chain Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Responsible Party: Charles Hesdorffer, MD, Columbia University
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/15927; CPMC-IRB-9041; CPMC-CAMP-009A
Record Dates: First submitted 2001-06-06; First posted 2001-06-06 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Amyloidosis
Keywords: amyloidosis; arthritis & connective tissue diseases; genetic diseases and dysmorphic syndromes; hematopoietic/lymphoid cancer; oncologic disorders; plasma cell neoplasm; primary systemic amyloidosis; rare disease
MeSH Terms: conditions — Amyloidosis; Arthritis; Connective Tissue Diseases; Genetic Diseases, Inborn; Hematologic Neoplasms; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis; Rare Diseases | interventions — Melphalan

INTERVENTIONS:
Drug: Melphalan — 100 mg/m2 twice a day from Days -2 and -1 as induction therapy
Procedure: Autologous Stem Cell Transplantation — Bone marrow and peripheral blood stem cells harvested

SUMMARY:
OBJECTIVES: I. Determine the response, disease-free survival, and overall survival of patients with primary light chain amyloidosis treated with high-dose melphalan and autologous stem cell transplantation.

II. Determine the toxicity of this regimen in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients may receive induction chemotherapy before study entry. Patients then receive filgrastim (G-CSF) or another growth factor for 4-6 days as peripheral blood stem cell (PBSC) mobilization. PBSC (or bone marrow) is harvested over 2-3 days.

Patients receive high-dose melphalan IV over 30 minutes twice daily on days -2 and -1. PBSC and/or bone marrow is reinfused on day 0. Patients receive G-CSF beginning on day 0 and continuing until blood counts recover. This course may be repeated 4-12 weeks later.

Patients are followed every 3 months for 1 year and then annually for 5 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

Disease Characteristics

* Histologically confirmed primary amyloidosis
* Ineligible for other high priority national or international study

Prior/Concurrent Therapy

* Biologic therapy: Concurrent participation in gene therapy trials allowed
* Chemotherapy: Prior chemotherapy allowed No other concurrent chemotherapy
* Endocrine therapy: No concurrent steroids unless given with amphotericin B, for adrenal failure, or for septic shock No concurrent hormones except for non-disease-related conditions (e.g., insulin for diabetes)
* Other: No concurrent barbiturates or acetaminophen Concurrent participation in supportive care trials allowed

Patient Characteristics

* Performance status: ECOG 0-3
* Hepatic: Bilirubin less than 2 times normal
* Renal: Creatinine less than 2.5 mg/dL OR On stable hemodialysis
* Pulmonary: DLCO at least 60% predicted OR Clearance by pulmonologist
* Other: HIV negative

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 1999-07; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Response, disease-free survial, and overall survial; response will be determined by the change in organ dysfunction

SECONDARY OUTCOMES:
Toxicity of high dose chemotherapy regimen

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Hesdorffer, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States